CLINICAL TRIAL: NCT06632015
Title: The Effects of Calcium Hydroxide and Diclofenac Sodium on Post-Endodontic Pain: A Double-Blinded, Parallel Group, Randomized Controlled Clinical Trial
Brief Title: Effect of DCS on Post-Endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, BÜŞRA FİDANOĞLU, Research Assistant, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMKU-001
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Post Endodontic Pain
Keywords: Endodontics; Post-Endodontic Pain; Calcium Hydroxide; Diclofenac Sodium; Intracanal Medicament; Randomized Controlled Trial
MeSH Terms: interventions — Calcium Hydroxide; Diclofenac; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calcium Hydroxide (CH) (Experimental): Working length was determined using a size 15 K-file and an apex locator (Morita Root ZX, Tokyo, Japan) and confirmed radiographically. Chemomechanical preparation was performed as described in the protocol. After drying with paper points, 1 mL of distilled water mixed with 1 g calcium hydroxide powder was placed as the intracanal medicament.
  Interventions: Drug: Calcium Hydroxide (CH)
- Diclofenac Sodium (DCS) (Experimental): Procedures as in Arm 1. After drying with paper points, 1 mL of distilled water mixed with 1 g diclofenac sodium powder was placed as the intracanal medicament.
  Interventions: Drug: Diclofenac Sodium (DCS)
- Calcium Hydroxide + Diclofenac Sodium (CH+DCS) (Experimental): Procedures as in Arm 1. After drying with paper points, 1 mL of distilled water mixed with 950 mg calcium hydroxide powder and 50 mg diclofenac sodium powder was placed as the intracanal medicament.
  Interventions: Drug: Calcium Hydroxide + Diclofenac Sodium (CH + DCS)

INTERVENTIONS:
Drug: Calcium Hydroxide (CH) — 1 mL distilled water mixed with 1 g calcium hydroxide powder, placed into the root canals using a lentulo spiral.
  Arms: Calcium Hydroxide (CH)
Drug: Diclofenac Sodium (DCS) — 1 mL distilled water mixed with 1 g diclofenac sodium powder, placed into the root canals using a lentulo spiral.
  Arms: Diclofenac Sodium (DCS)
Drug: Calcium Hydroxide + Diclofenac Sodium (CH + DCS) — 1 mL distilled water mixed with 950 mg calcium hydroxide powder and 50 mg diclofenac sodium powder, placed into the root canals using a lentulo spiral.
  Arms: Calcium Hydroxide + Diclofenac Sodium (CH+DCS)

SUMMARY:
The aim of this randomized, triple-blind, parallel-group clinical trial was to evaluate the effects of calcium hydroxide (CH), diclofenac sodium (DCS), and their combination (CH+DCS) as intracanal medicaments on post-endodontic pain in mandibular molars diagnosed with symptomatic apical periodontitis. Ninety patients were randomly assigned to three groups (CH, DCS, or CH+DCS; n=30 each). Pain intensity was recorded using a 100 mm Visual Analog Scale (VAS) over 7 days following treatment, and the number of analgesic tablets taken was also recorded. Statistical analyses were performed using Kruskal-Wallis, Friedman, Wilcoxon signed-rank, and Chi-square tests, with significance set at 0.05. The null hypothesis stated that there would be no significant difference in post-endodontic pain among the groups.

DETAILED DESCRIPTION:
This randomized, triple-blind, parallel-group clinical trial included 90 patients aged 18-60 years with a single mandibular molar diagnosed with symptomatic apical periodontitis. Sample size was calculated based on a priori power analysis to detect significant differences in post-endodontic pain, resulting in 30 participants per group.

All endodontic procedures were performed by a single clinician under local anesthesia. After tooth isolation and access cavity preparation, working length was determined using K-files and an apex locator, verified radiographically. Chemomechanical preparation was performed using Reciproc files according to canal dimensions. Irrigation was performed using 2.5% NaOCl and 17% EDTA, followed by canal drying.

Patients were randomly assigned to three groups according to the intracanal medicament:

Group 1 (CH): 1 g Calcium Hydroxide mixed with 1 mL distilled water Group 2 (DCS): 1 g Diclofenac Sodium mixed with 1 mL distilled water Group 3 (CH + DCS): 950 mg Calcium Hydroxide + 50 mg Diclofenac Sodium mixed with 1 mL distilled water The canals were sealed temporarily. Postoperative pain was recorded daily for 7 days using a 100 mm Visual Analog Scale (VAS). Patients also recorded the number of analgesic tablets taken. Pain assessments were conducted by a blinded researcher. For pain management, 400 mg ibuprofen was prescribed if needed, with contact support provided for severe pain.

At the second session, medicaments were removed, final irrigation was performed, canals were dried, and obturation was completed using a single-cone technique with gutta-percha and calcium silicate sealer. Teeth were restored with resin composite.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Systemically healthy (ASA I-II)
* Diagnosed with symptomatic irreversible pulpitis or symptomatic apical periodontitis in mandibular molars (characterized by spontaneous pain or prolonged pain in response to cold test, and presence of percussion sensitivity)
* Positive response to Electric Pulp Testing (EPT) and cold testing
* Periapical Index (PAI) score of 1 or 2 according to Ørstavik et al. (1986)
* Pre-operative pain level ≥50 mm on the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 100 (most severe pain)

Exclusion Criteria:

* History of psychiatric disorders
* Allergic reactions
* Pregnancy
* Use of analgesics within the previous 24 hours
* Use of antibiotics within the last 3 months
* Teeth with a sinus tract or history of abscess formation
* Periodontal pocket depth >3 mm
* Root resorption, root fractures, or ankylosis
* Previous root canal treatment on the selected tooth
* Teeth requiring prosthetic restoration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Post-Endodontic Pain | Baseline and Days 1-7 post-treatment
  Pre-operative (before treatment) and post-operative pain were assessed using the Visual Analog Scale (VAS), a 100 mm horizontal line with numerical values. Patients rated their pain on the VAS, and pain severity was categorized as follows: No pain (0 mm), mild pain (1-19 mm), moderate pain (20-49 mm), severe pain (50-79 mm), and very severe pain (80-100 mm). Post-operative pain measurements were taken on Days 1, 2, 3, 4, 5, 6, and 7 after intracanal medicament application.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect patient privacy and confidentiality.

REFERENCES:
- [Derived] Fidanoglu B, Tufenkci P, Sari M. The effects of calcium hydroxide and diclofenac sodium as root canal medicaments on post-endodontic pain: a double-blinded, parallel group, randomized controlled clinical trial. Odontology. 2025 Nov 9. doi: 10.1007/s10266-025-01252-9. Online ahead of print. PMID 41206809